CLINICAL TRIAL: NCT05168111
Title: The Correlation Between the Metabolism and the Functional Status of Multiple Organs in the Early Stage of Diquat Poisoning---A Multicenter Observational Study
Brief Title: The Correlation Between the Metabolism and the Functional Status of Multiple Organs in the Early Stage of Diquat Poisoning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1068
Record Dates: First submitted 2021-12-15; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Diquat Poisoning
Keywords: Diquat Metabolomics Toxicology Multicenter

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients of Diquat poisoning
  Interventions: Diagnostic Test: Detect the serum sample
- normal persons
  Interventions: Diagnostic Test: Detect the serum sample

INTERVENTIONS:
Diagnostic Test: Detect the serum sample — Detect the serum sample

SUMMARY:
Diquat (DQ), as a conductive biocidal herbicide, is classified as medium according to Chinese pesticide toxicity classification standards. Since the sale and use of paraquat are stopped in 2016, incidents of diquat poisoning have begun to increase. Diquat is very toxic to the human body. Mistake of Diquat can cause damage to multiple organs throughout the body. It has a high fatality rate and no specific treatment.The treatment method has become a research hotspot of modern poisoning treatment.

The degree of organ dysfunction caused by DQ poisoning is mainly related to the patient's intake and the distribution of the poison in the human body.So far, the distribution concentration of DQ under the influence of the time gradient in the body and the influence of DQ on the human environment，metabolimics,，immune regulation activity and the comprehensive mechanism of action of various inflammatory factors have not been fully elucidated. Therefore, this research mainly focuses on analyzing the internal environment metabolism research in patients with DQ poisoning, and to conduct exploratory research on the severity of the impact on their organ functions

ELIGIBILITY:
Inclusion Criteria:

1.Time from poisoning to hospital admission: within 6 hours, 2 The age is greater than 18 years old, less than 65 years old 3 There is at least one target organ dysfunction 4 Previous physical fitness 5 No bad habits (drug use, alcohol addiction)

Exclusion Criteria:

1. Refuse to join this study
2. Missing/incomplete information
3. Pregnant women, vulnerable groups such as those who have no capacity for civil conduct and cannot determine the consent of their attorneys
4. Chronic organ dysfunction (chronic heart insufficiency, chronic respiratory insufficiency, chronic renal insufficiency, chronic Liver insufficiency)
5. Tumors, blood system diseases, various systemic immune diseases
6. Various infectious diseases (various hepatitis, tuberculosis, AIDS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute poisoning of diquat are mainly selected.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The poison metabolomics of Diquat | 2022-06
  Improve the correlation between the concentration and metabolism rate of diquat poisoning in vivo and metabolomics and the co-damage color of body organs for bioinformatics analysis and summary

CONTACTS AND LOCATIONS:
Overall Officials: Yongan Xu, Study Director — SAHZU
Locations (1):
- SAHZU, Hanzhou, Zhejiang, China